CLINICAL TRIAL: NCT02264613
Title: A Phase 1/2a Open-Label Study to Determine the Safety and Tolerability of ALRN-6924 Alone or in Combination in Patients With Advanced Solid Tumors or Lymphomas Expressing Wild-Type p53 Protein
Brief Title: ALRN-6924 in Patients With Advanced Solid Tumors or Lymphomas
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Aileron Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALRN-6924-1-01
Record Dates: First submitted 2014-10-07; First posted 2014-10-15 (Estimated); Results first posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumor; Lymphoma; Peripheral T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Regimen A (DR-A) (Experimental): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle.
  Interventions: Drug: ALRN-6924
- Dose Regimen B (DR-B) (Experimental): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 4, 8 and 11 of a 21-day cycle
  Interventions: Drug: ALRN-6924
- Dose Regimen C (DR-C) (Experimental): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 3 and 5 of a 21-day cycle
  Interventions: Drug: ALRN-6924
- Combination with palbociclib (Experimental): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle Drug: Palbociclib Fixed-dose capsule administered orally on days 1 through 21 of a 28-day cycle
  Interventions: Drug: ALRN-6924

INTERVENTIONS:
Drug: ALRN-6924 — ALRN-6924 will be administered as an IV infusion

SUMMARY:
This study evaluates the anti-tumor effects of ALRN-6924 in patients with advanced solid tumors or lymphomas with WT TP53.

DETAILED DESCRIPTION:
Open label, multi center, Phase 1 (dose escalation) and Phase 2a (dose expansion) study design to evaluate safety, tolerability, PK, PD and anti-tumor effects of ALRN-6924, alone or in combination with palbociclib, in patients with advanced solid tumors or lymphomas with wild-type (WT) TP53. ALRN-6924 is a stabilized cell-permeating peptide designed to disrupt the interaction between the p53 tumor suppressor protein and its predominant endogenous inhibitors, murine double minute 2 (MDM2) and murine double minute X (MDMX).

The Phase 1 portion of the study will enroll adults with histologically or cytologically confirmed malignancies that are metastatic or unresectable and for which standard treatment(s) are not available or are no longer effective. The Phase 2a portion of the study consists of separate cohorts that will enroll distinct groups of patients with specific solid tumors and/or lymphomas to further investigate the clinical safety profile and potential efficacy of ALRN-6924 alone or in a combination regimen.

Treatment will continue until unacceptable toxicity, patient or physician decision to discontinue therapy or disease progression that is either symptomatic, rapidly progressive, requires urgent intervention or is associated with a decline in performance status.

Patients with PTCL have been selected as a group to be further studied in Phase 2a.

Patients with MDM2-amplified or MDM2/CDK4-co-amplified solid tumors have been selected as another group to be further studied in Phase 2a.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed solid tumor or lymphoma that is not amenable to standard therapies.
* Cohort specific biomarkers, including confirmed or anticipated WT TP53 (Phase 1 and PTCL expansion cohorts) and MDM2-amplification or MDM2/CDK4-co-amplification (solid tumor expansion cohort)
* At least one target lesion that is measurable by RECIST 1.1, RANO or IWG 2014, as appropriate for tumor type
* ECOG (Eastern Cooperative Oncology Group) performance status 0-1
* Adequate coagulation and hematologic function
* Adequate hepatic and renal function
* Sufficient wash out from prior therapies and recovery from all significant acute toxicities

Key Exclusion Criteria

* Prior treatment with an MDM2 inhibitor, with protocol specified exceptions
* Known hypersensitivity to any study drug component
* Protocol specified cardiovascular risk factors
* Clinically significant gastrointestinal bleeding within 6 months
* Clinically significant third-space fluid accumulation
* Active uncontrolled infection, including HIV/AIDS or Hepatitis B or C
* HPV positive tumors
* Second malignancy within two years, with protocol specified exceptions
* Pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Birmingham, Alabama
  - Duarte, California
  - Denver, Colorado
  - Sarasota, Florida
  - Tampa, Florida
  - Boston, Massachusetts
  - New York, New York
  - The Bronx, New York
  - Greenville, South Carolina
  - Nashville, Tennessee
  - Houston, Texas
  - Seattle, Washington

REFERENCES:
- [Derived] Zhou X, Singh M, Sanz Santos G, Guerlavais V, Carvajal LA, Aivado M, Zhan Y, Oliveira MMS, Westerberg LS, Annis DA, Johnsen JI, Selivanova G. Pharmacologic Activation of p53 Triggers Viral Mimicry Response Thereby Abolishing Tumor Immune Evasion and Promoting Antitumor Immunity. Cancer Discov. 2021 Dec 1;11(12):3090-3105. doi: 10.1158/2159-8290.CD-20-1741. PMID 34230007

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Regimen A (DR-A) Escalation (0.16 mg/kg); Dose Regimen A (DR-A) Escalation (0.32 mg/kg); Dose Regimen A (DR-A) Escalation (0.64 mg/kg); Dose Regimen A (DR-A) Escalation (1.25 mg/kg); Dose Regimen A (DR-A) Escalation (2.10 mg/kg); Dose Regiment A (DR-A) Escalation (3.10 mg/kg); Dose Regimen A (DR-A) Escalation (4.40 mg/kg); Dose Regimen B (DR-B) Escalation (0.53 mg/kg); Dose Regimen B (DR-B) Escalation (0.80 mg/kg); Dose Regimen B (DR-B) Escalation (1.10 mg/kg); Dose Regimen B (DR-B) Escalation (1.50 mg/kg); Dose Regimen B (DR-B) Escalation (2.00 mg/kg); Dose Regimen B (DR-B) Escalation (2.70 mg/kg); Dose Regimen A (DR-A) PTCL Expansion: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle.
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Dose Regimen B (DR-B) Escalation (0.32 mg/kg): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 4, 8 and 11 of a 21-day cycle
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Dose Regimen C (DR-C) PTCL Expansion: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 3 and 5 of a 21-day cycle
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Combination With Palbociclib Expansion: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle Drug: Palbociclib Fixed-dose capsule administered orally on days 1 through 21 of a 28-day cycle
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
Period: Overall Study
Arm/Group | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) | Dose Regimen A (DR-A) Escalation (2.10 mg/kg) | Dose Regiment A (DR-A) Escalation (3.10 mg/kg) | Dose Regimen A (DR-A) Escalation (4.40 mg/kg) | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) | Dose Regimen B (DR-B) Escalation (0.80 mg/kg) | Dose Regimen B (DR-B) Escalation (1.10 mg/kg) | Dose Regimen B (DR-B) Escalation (1.50 mg/kg) | Dose Regimen B (DR-B) Escalation (2.00 mg/kg) | Dose Regimen B (DR-B) Escalation (2.70 mg/kg) | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion | Combination With Palbociclib Expansion
Started | 5 | 3 | 4 | 3 | 6 | 9 | 11 | 3 | 5 | 3 | 4 | 4 | 5 | 6 | 21 | 16 | 34
Completed | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 7
Not Completed | 5 | 3 | 4 | 2 | 5 | 9 | 10 | 3 | 5 | 3 | 4 | 4 | 5 | 4 | 20 | 16 | 27

BASELINE CHARACTERISTICS:
Groups:
- Dose Regimen A (DR-A) Escalation (3.10 mg/kg); Dose Regimen A (DR-A) Escalation (4.40 mg/kg); Dose Regimen A (DR-A) PTCL Expansion: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle.
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Dose Regimen B (DR-B) Escalation (0.53 mg/kg); Dose Regimen B (DR-B) Escalation (0.80 mg/kg); Dose Regimen B (DR-B) Escalation (1.10 mg/kg); Dose Regimen B (DR-B) Escalation (1.50 mg/kg); Dose Regimen B (DR-B) Escalation (2.00 mg/kg); Dose Regimen B (DR-B) Escalation (2.70 mg/kg): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 4, 8 and 11 of a 21-day cycle
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Total: Total of all reporting groups
Arm/Group | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) | Dose Regimen A (DR-A) Escalation (2.10 mg/kg) | Dose Regimen A (DR-A) Escalation (3.10 mg/kg) | Dose Regimen A (DR-A) Escalation (4.40 mg/kg) | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) | Dose Regimen B (DR-B) Escalation (0.80 mg/kg) | Dose Regimen B (DR-B) Escalation (1.10 mg/kg) | Dose Regimen B (DR-B) Escalation (1.50 mg/kg) | Dose Regimen B (DR-B) Escalation (2.00 mg/kg) | Dose Regimen B (DR-B) Escalation (2.70 mg/kg) | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion | Combination With Palbociclib Expansion | Total
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6 | 9 | 11 | 3 | 5 | 3 | 4 | 4 | 5 | 6 | 21 | 16 | 34 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (15.04) | 50.7 (22.37) | 64.0 (5.29) | 66.3 (9.02) | 53.8 (13.75) | 59.3 (13.17) | 61.5 (11.01) | 58.9 (12.75) | 58.4 (12.76) | 54.7 (4.04) | 65.2 (8.64) | 55.3 (1.53) | 56.0 (17.78) | 49.3 (14.97) | 59.8 (16.62) | 59.5 (14.21) | 58.7 (11.77) | 58.5 (13.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 4 | 4 | 6 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 12 | 8 | 19 | 75
  Male | 3 | 1 | 2 | 2 | 2 | 5 | 5 | 0 | 3 | 1 | 2 | 2 | 3 | 4 | 9 | 8 | 15 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 4 | 12
  Not Hispanic or Latino | 4 | 3 | 2 | 2 | 5 | 7 | 11 | 2 | 3 | 3 | 4 | 4 | 5 | 5 | 18 | 12 | 30 | 120
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 1 | 0 | 2 | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 6 | 5 | 3 | 27
  White | 4 | 1 | 2 | 2 | 4 | 7 | 8 | 2 | 4 | 3 | 3 | 3 | 5 | 5 | 12 | 8 | 28 | 101
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 4 | 3 | 6 | 9 | 11 | 3 | 5 | 3 | 4 | 4 | 5 | 6 | 21 | 16 | 34 | 142

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Safety and Tolerability of ALRN-6924 in Adult Patients With Advanced Solid Tumors or Lymphomas With Wild-type (WT) TP53 Who Are Refractory to or Intolerant of Standard Therapy, or for Whom no Standard Therapy Exists
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v.4.0
Time Frame: From Day 1 of treatment until 30 days after the last cycle of treatment (each cycle in DR-A is 28 days, DR-B and DR-C is 21 days), an average of 138 Days
Measure: Count of Participants; unit: Participants
Groups:
- Dose Regimen A (DR-A) Escalation (1.25 mg/kg) Escalation; Dose Regimen A (DR-A) Escalation (2.10 mg/kg) Escalation; Dose Regimen A (DR-A) Escalation (3.10 mg/kg) Escalation; Dose Regimen A (DR-A) Escalation (4.40 mg/kg) Escalation; Dose Regimen A (DR-A) PTCL Expansion: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle.
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Combination With Palbociclib Expansion (DR-A): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle Drug: Palbociclib Fixed-dose capsule administered orally on days 1 through 21 of a 28-day cycle
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
Arm/Group | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) Escalation | Dose Regimen A (DR-A) Escalation (2.10 mg/kg) Escalation | Dose Regimen A (DR-A) Escalation (3.10 mg/kg) Escalation | Dose Regimen A (DR-A) Escalation (4.40 mg/kg) Escalation | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) | Dose Regimen B (DR-B) Escalation (0.80 mg/kg) | Dose Regimen B (DR-B) Escalation (1.10 mg/kg) | Dose Regimen B (DR-B) Escalation (1.50 mg/kg) | Dose Regimen B (DR-B) Escalation (2.00 mg/kg) | Dose Regimen B (DR-B) Escalation (2.70 mg/kg) | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion | Combination With Palbociclib Expansion (DR-A)
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6 | 9 | 11 | 3 | 5 | 3 | 4 | 4 | 5 | 6 | 21 | 16 | 34
Participants | 5 | 3 | 4 | 3 | 6 | 9 | 11 | 3 | 5 | 3 | 4 | 4 | 5 | 6 | 21 | 16 | 34

2. Primary Outcome: Evaluate the Safety and Tolerability of ALRN-6924 in Adult Patients With Advanced Solid Tumors or Lymphomas With Wild-type (WT) TP53 Who Are Refractory to or Intolerant of Standard Therapy, or for Whom no Standard Therapy Exists, Expansion
Description: Number of participants with treatment-related adverse events as assessed by CTCAE v.4.0
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion | Combination With Palbociclib Expansion (DR-A)
Number analyzed (Participants) | 21 | 16 | 34
Participants | 21 | 16 | 34

3. Primary Outcome: Determine the Maximum Tolerated Dose (MTD) of ALRN-6924 in Adult Patients With Advanced Solid Tumors or Lymphomas
Description: Determine the maximum tolerated dose (MTD)
Time Frame: as for outcome 1
Measure: Number; unit: mg/kg
Groups:
- Dose Regimen A (DR-A) Escalation: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle.
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Dose Regimen B (DR-B) Escalation: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 4, 8 and 11 of a 21-day cycle
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
Arm/Group | Dose Regimen A (DR-A) Escalation | Dose Regimen B (DR-B) Escalation
Number analyzed (Participants) | 41 | 30
mg/kg | 3.1 | NA — No MTD found

4. Primary Outcome: Determine Overall Response Rate
Description: The proportion of efficacy-evaluable patients who achieve complete response (CR) or partial response (PR), per investigator assessment, in accordance with RECIST 1.1 or iRECIST (for solid tumor patients) or Response Assessment in Neuro-Oncology (RANO) criteria (for glioblastoma patients).
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion
Number analyzed (Participants) | 21 | 16
Participants | 2 | 2

5. Secondary Outcome: Assess Additional Measures of Anti-tumor Activity, Including Duration of Response, Progression Free Survival, Overall Survival and Time to Response
Description: as for outcome 4
Time Frame: as for outcome 1
Population: The efficacy evaluable population was defined as those patients who met all of the following criteria: (1) Received at least 1 dose of ALRN-6924 at a dose level at least 0.8 mg/kg per infusion (2) Had at least 1 postbaseline evaluation or had clinical disease progression (3) Were TP53 wild type or indeterminate (as assessed by the central laboratory; if not assessed by central laboratory, as assessed by the local laboratory.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) | Dose Regimen A (DR-A) Escalation (2.10 mg/kg) | Dose Regimen A (DR-A) Escalation (3.10 mg/kg) | Dose Regimen A (DR-A) Escalation (4.40 mg/kg) | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) | Dose Regimen B (DR-B) Escalation (0.80 mg/kg) | Dose Regimen B (DR-B) Escalation (1.10 mg/kg) | Dose Regimen B (DR-B) Escalation (1.50 mg/kg) | Dose Regimen B (DR-B) Escalation (2.00 mg/kg) | Dose Regimen B (DR-B) Escalation (2.70 mg/kg) | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion | Combination With Palbociclib Expansion
Number analyzed (Participants) | 0 | 0 | 0 | 2 | 3 | 7 | 8 | 0 | 0 | 3 | 4 | 4 | 4 | 6 | 16 | 11 | 25
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0

6. Secondary Outcome: Determine Pharmacokinetic Parameters of ALRN-6924 When Administered to Patients With Advanced Solid Tumors or Lymphomas
Description: Time of Peak Plasma Concentration (Tmax)
Time Frame: 8 weeks
Population: The Pharmacokinetic Analysis Population included all subjects who received at least one dose of ALRN-6924 with sufficient plasma sample data to assess PK parameters, and with no major protocol violations. Plasma samples for subjects in the Combination With Palbociclib Expansion arm were collected but will not be processed or analyzed due to a protocol-level decision for this expansion arm to discontinue pharmacokinetic data collection.
Measure: Median (Full Range); unit: hour
Arm/Group | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) Escalation | Dose Regimen A (DR-A) Escalation (2.10 mg/kg) Escalation | Dose Regimen A (DR-A) Escalation (3.10 mg/kg) Escalation | Dose Regimen A (DR-A) Escalation (4.40 mg/kg) Escalation | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) | Dose Regimen B (DR-B) Escalation (0.80 mg/kg) | Dose Regimen B (DR-B) Escalation (1.10 mg/kg) | Dose Regimen B (DR-B) Escalation (1.50 mg/kg) | Dose Regimen B (DR-B) Escalation (2.00 mg/kg) | Dose Regimen B (DR-B) Escalation (2.70 mg/kg) | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion | Combination With Palbociclib Expansion
Number analyzed (Participants) | 5 | 3 | 4 | 3 | 6 | 9 | 11 | 3 | 5 | 3 | 4 | 4 | 5 | 6 | 21 | 16 | 0
hour | 0.03 [0.00 to 0.52] | 0.13 [0.07 to 0.50] | 0.04 [0.02 to 0.47] | 0.04 [0.02 to 0.07] | 0.29 [0.00 to 1.00] | 0.12 [0.00 to 0.65] | 0.06 [0.03 to 1.00] | 0.17 [0.15 to 0.18] | 0.22 [0.02 to 1.00] | 0.08 [0.07 to 0.08] | 0.29 [0.02 to 0.50] | 0.08 [0.02 to 1.00] | 0.30 [0.05 to 0.50] | 0.03 [0.00 to 1.02] | 0.05 [0.02 to 0.48] | 0.05 [0.00 to 0.52] |

ADVERSE EVENTS:
Time Frame: From Day 1 of treatment until the last post treatment visit 30 days after the last treatment dose, an average of 138 Days
Groups:
- Dose Regimen A (DR-A) Escalation (2.1 mg/kg); Dose Regimen A (DR-A) Escalation (3.1 mg/kg); Dose Regimen A (DR-A) Escalation (4.4 mg/kg); Dose Regimen A (DR-A) PTCL Expansion: Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 8 and 15 of a 28-day cycle.
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
- Dose Regimen B (DR-B) Escalation (0.8 mg/kg); Dose Regimen B (DR-B) Escalation (1.1 mg/kg); Dose Regimen B (DR-B) Escalation (1.5 mg/kg); Dose Regimen B (DR-B) Escalation (2.0 mg/kg); Dose Regimen B (DR-B) Escalation (2.7 mg/kg): Drug: ALRN-6924 Weight-based-dosing administered IV on days 1, 4, 8 and 11 of a 21-day cycle
  ALRN-6924: ALRN-6924 will be administered as an IV infusion
Arm/Group | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) | Dose Regimen A (DR-A) Escalation (2.1 mg/kg) | Dose Regimen A (DR-A) Escalation (3.1 mg/kg) | Dose Regimen A (DR-A) Escalation (4.4 mg/kg) | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) | Dose Regimen B (DR-B) Escalation (0.8 mg/kg) | Dose Regimen B (DR-B) Escalation (1.1 mg/kg) | Dose Regimen B (DR-B) Escalation (1.5 mg/kg) | Dose Regimen B (DR-B) Escalation (2.0 mg/kg) | Dose Regimen B (DR-B) Escalation (2.7 mg/kg) | Dose Regimen A (DR-A) PTCL Expansion | Dose Regimen C (DR-C) PTCL Expansion | Combination With Palbociclib Expansion
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/3 | 0/4 | 0/3 | 0/6 | 0/9 | 0/11 | 0/3 | 0/5 | 0/3 | 0/4 | 0/4 | 0/5 | 0/6 | 0/21 | 0/16 | 5/34
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/3 | 0/4 | 1/3 | 0/6 | 2/9 | 4/11 | 0/3 | 1/5 | 0/3 | 0/4 | 0/4 | 0/5 | 0/6 | 7/21 | 7/16 | 5/34
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 4/4 | 3/3 | 6/6 | 9/9 | 11/11 | 3/3 | 5/5 | 3/3 | 4/4 | 4/4 | 5/5 | 6/6 | 19/21 | 15/16 | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) (N=5) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) (N=3) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) (N=4) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) (N=3) | Dose Regimen A (DR-A) Escalation (2.1 mg/kg) (N=6) | Dose Regimen A (DR-A) Escalation (3.1 mg/kg) (N=9) | Dose Regimen A (DR-A) Escalation (4.4 mg/kg) (N=11) | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) (N=3) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) (N=5) | Dose Regimen B (DR-B) Escalation (0.8 mg/kg) (N=3) | Dose Regimen B (DR-B) Escalation (1.1 mg/kg) (N=4) | Dose Regimen B (DR-B) Escalation (1.5 mg/kg) (N=4) | Dose Regimen B (DR-B) Escalation (2.0 mg/kg) (N=5) | Dose Regimen B (DR-B) Escalation (2.7 mg/kg) (N=6) | Dose Regimen A (DR-A) PTCL Expansion (N=21) | Dose Regimen C (DR-C) PTCL Expansion (N=16) | Combination With Palbociclib Expansion (N=34)
hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AKI (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
hypercalcemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
CDIFF (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Histiocytosis Hamatophagic (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hypokalemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperbilirubinemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrulation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Escherichia bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CVA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal bacteremia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue Hemorrhage (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose Regimen A (DR-A) Escalation (0.16 mg/kg) (N=5) | Dose Regimen A (DR-A) Escalation (0.32 mg/kg) (N=3) | Dose Regimen A (DR-A) Escalation (0.64 mg/kg) (N=4) | Dose Regimen A (DR-A) Escalation (1.25 mg/kg) (N=3) | Dose Regimen A (DR-A) Escalation (2.1 mg/kg) (N=6) | Dose Regimen A (DR-A) Escalation (3.1 mg/kg) (N=9) | Dose Regimen A (DR-A) Escalation (4.4 mg/kg) (N=11) | Dose Regimen B (DR-B) Escalation (0.32 mg/kg) (N=3) | Dose Regimen B (DR-B) Escalation (0.53 mg/kg) (N=5) | Dose Regimen B (DR-B) Escalation (0.8 mg/kg) (N=3) | Dose Regimen B (DR-B) Escalation (1.1 mg/kg) (N=4) | Dose Regimen B (DR-B) Escalation (1.5 mg/kg) (N=4) | Dose Regimen B (DR-B) Escalation (2.0 mg/kg) (N=5) | Dose Regimen B (DR-B) Escalation (2.7 mg/kg) (N=6) | Dose Regimen A (DR-A) PTCL Expansion (N=21) | Dose Regimen C (DR-C) PTCL Expansion (N=16) | Combination With Palbociclib Expansion (N=34)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 9 (9) | 6 (6) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 4 (4) | 5 (5) | 3 (3) | 10 (10) | 7 (7) | 19 (19)
Vomitting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4) | 7 (7) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 13 (13)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 7 (7)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0) | 2 (2) | 3 (3) | 5 (5) | 4 (4) | 9 (9) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 2 (2) | 9 (9) | 6 (6) | 12 (12)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 2 (2) | 4 (4) | 4 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 1 (1) | 7 (7)
thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 12 (12)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 24 (24)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 12 (12)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4)
Hyperbilirubinemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/13/NCT02264613/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/13/NCT02264613/SAP_001.pdf